CLINICAL TRIAL: NCT07227324
Title: Cannabis Use Registry to Improve Overall Understanding of Symptoms (CURIOUS)
Acronym: CURIOUS
Status: Recruiting | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Ontracka (Unknown)
Responsible Party: Sponsor
Other Study IDs: A24-181
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use; Cancer
Keywords: cannabis; cancer; symptom management; education
MeSH Terms: conditions — Neoplasms; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through partnership with Ontracka, the HealthPartners Institute Cancer Research Center created a secure and compliant app-based technology with the ability to seamlessly collect patient-level data on symptoms, cannabis use, real-time response to cannabis consumption, and patient-reported changes in supportive care medications such as opioids and antiemetics. By joining this registry, patients will have access to expert cannabis education, dosing recommendations, and easy symptom tracking. Patients with cancer and their oncology clinicians can utilize this reliable, cancer-specific data to help them make informed decisions together about how cannabis could be incorporated into a treatment plan. To learn more and sign up, visit https://study.ontracka.com/cannabiscurious

DETAILED DESCRIPTION:
The CURIOUS project enhances the ability to seamlessly collect patient-level data on symptoms, cannabis use, real-time response to cannabis consumption, and patient-reported changes in supportive care medications such as opioids and antiemetics. Any patient interested in cannabis use can access the weblink to receive information about the CURIOUS study. An electronic version of the informed consent document will be available for them to review.

Patients interested in participating in the CURIOUS study will sign an electronic consent form on the app that describes how data will be used and stored by the HealthPartners and the Ontracka teams. They will be required to submit their name, email, and date of birth. This will automatically establish an account in the OnTracka platform and provide instruction on how to download and install the OnTracka mobile app. After patients consent to participate, they will receive access to the Ontracka app to track cannabis consumption and symptom responses as well as complete embedded validated questionnaires sent to them through the app at defined intervals; NCI PRO-CTCAE (PRO) (every other week), PROMIS Global (QOL) (every 4 weeks) and medication logs (every 4 weeks) through 12 weeks. After week 12 collection, they will complete all surveys once again in month 6 and month 12.

ELIGIBILITY:
Inclusion Criteria:

* any adult aged 18 or older who is diagnosed with cancer and using cannabis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: any adult aged 18 or older who is diagnosed with cancer and using cannabis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Adherence | from enrollment to the first 90 days of study participation
  Assess adherence to CURIOUS platform by determining the percentage of consented patients who access the app/survey at least once per month during the first 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners Institute Cancer Research Center, Saint Louis Park, Minnesota, United States

REFERENCES:
- See also: Visit this link to learn more and sign up — https://study.ontracka.com/cannabiscurious